CLINICAL TRIAL: NCT06243796
Title: Seroma Formation After Modified Radical Mastectomy With Flap Fixation Technique in Breast Cancer Patients: Nakhon Phanom Hospital - a Single Blinded Randomized Control Trial
Brief Title: Seroma Formation After Modified Radical Mastectomy With Flap Fixation Technique in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nakhon Phanom Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 39/2566
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Results first posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: Breast-cancer
Keywords: Mastectomy flap fixation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Single blinded randomized control trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The statistician will generate randomization list from block randomization, then concealed envelope
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flap fixation (Experimental): After completing the modified radical mastectomy procedure, the researcher will use absorbable suture (vicryl), multiple alternating stitches 2.5 cm apart between the subcutaneous tissues of the skin flaps and the underlying muscles at various parts of the flap and also, at the wound edge.
  Interventions: Procedure: Flap fixation technique
- Non flap fixation (No Intervention): After mastectomy, the researcher will close the wound in the conventional method.

INTERVENTIONS:
Procedure: Flap fixation technique — After complete the modified radical mastectomy procedure, the researcher will use absorbable sutures (vicryl), multiple alternating stitched 2.5 cm apart between the subcutaneous of the flap and underlying muscle
  Arms: Flap fixation

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of mastectomy flap fixation in breast cancer patients. The main questions it aims to answer are:

- To compare seroma formation after mastectomy flap fixation with conventional surgery in breast cancer patients Participants will be randomly divided into 2 groups,

1. Mastectomy flap fixation
2. Conventional surgery with non flap fixation. Researchers will record the amount and color of drainage fluid, patient and tumor characteristics, and operative related factor after surgery.

Researchers will compare with conventional surgery to see if seroma formation, and wound infection.

DETAILED DESCRIPTION:
Seroma is collection of blood plasma or lymphatic fluid under skin flap or axillary dead space. It occurred after modified radical mastectomy. Patient will have subcutaneous swelling or edema which be confirmed by physical examination or bedside ultrasound. It categorized by common terminology criteria for adverse events version 5.0 for 3 grades.

1. asymptomatic
2. symptomatic with medical intervention or simple aspiration
3. symptomatic with required interventional radiology or operative intervention.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer (CA Breast) patients plan to modified radical mastectomy
* Operable case, or Resectable case

Exclusion Criteria:

* Having medical bleeding tendency e.g., Idiopathic Thrombocytopenia (ITP), leukemia, other bleeding disorder
* Immunocompromised e.g., HIV, Systemic Lupus Erythematosus (SLE), liver cirrhosis, immunosuppressive drug
* Other modified radical mastectomy whom required reconstruction, flap coverage e.g., Transverse Rectus Abdominis Musculocutaneous (TRAM) flap, Latissimus Dorsi (LD) flap
* Past history of mammoplasty, augmentation
* Past history of axillary lymphatic system operation
* Pregnant women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natawan Hunpayon, MD, Principal Investigator — Nakhon Phanom Hospital
Locations (1):
- Nakhon Phanom hospital, Nakhon Phanom, Thailand

IPD SHARING:
Plan to Share IPD: Yes
De-identify data
Supporting Information: Study Protocol, SAP
Time Frame: 1 year after publication for a period of 2 years
Access Criteria: Access to trial Individual Patient Data (IPD) can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of research proposal and statistical analysis plan (SAP) and execution of Data Sharing Agreement (DSA). For more information or to submit a request, please contact e-mail: sutthichain@gmail.com.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A single-blinded randomized control trial was conducted between December 2023 to June 2024. All operable breast cancer patients who were 18 years old and over, early and locally advance breast cancer who underwent modified radical mastectomy by single surgeon in Nakhonphanom hospital were screened
Pre-assignment Details: Excluded accidental finding liver cirrhosis before surgery (n=1), plan to move another province (n=1)
Groups:
- Flap Fixation (n=34): After completing the modified radical mastectomy procedure, the researcher will use absorbable suture (vicryl), multiple alternating stitches 2.5 cm apart between the subcutaneous tissues of the skin flaps and the underlying muscles at various parts of the flap and also, at the wound edge.
  Flap fixation technique: After complete the modified radical mastectomy procedure, the researcher will use absorbable sutures (vicryl), multiple alternating stitched 2.5 cm apart between the subcutaneous of the flap and underlying muscle
- Non Flap Fixation (n=34): After mastectomy, the researcher will close the wound in the conventional method.
Period: Overall Study
Arm/Group | Flap Fixation (n=34) | Non Flap Fixation (n=34)
Started | 34 | 34
Completed | 34 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Flap Fixation: Average age was 53±14 years. 13 patients with class I obesity (BMI > 25kg/m2) and above. 5 (14.7%)patients received neoadjuvant chemotherapy. Average operative time were 57±10 minutes. Average blood loss was 33.53±13.23 ml.
  Most of breast cancer cell type in this group was invasive ductal carcinoma = 32. Average tumor size in group A was 3.5 cm. Most of patients in this group were diagnosed in stage 2A, 14(41.18%).1 patients had distance metastasis, (2.94%).
- Non Flap Fixation: Average 58±10 years. 13 patients with class I obesity (BMI > 25kg/m2) and above. 9 (26.47%) patients received neoadjuvant chemotherapy. Average operative time was 58±10 minutes. Average blood loss was 35.88±17.60 ml.
  Most of breast cancer cell type in this group was invasive ductal carcinoma = 31 Average tumor size 4.09 cm. Most of patients in this group were diagnosed in stage 2A, 12 (35.29%). 4 (11.76%) patients had distance metastasis.
- Total: Total of all reporting groups
Arm/Group | Flap Fixation | Non Flap Fixation | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] — Age in years, Continuous
  years | 53 (24) | 58 (10) | 56 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 34 | 68
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 34 | 34 | 68
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Nakhon Phanom hospital, Thailand
  participants
    Thailand | 34 | 34 | 68
Co-morbidity [Count of Participants; unit: Participants] — Had one or more underlying medical conditions
  Participants | 18 | 22 | 40
Body mass index [Mean (Standard Deviation); unit: kg/m2] — Body mass index (Body weight)kg/(Height)m2
  kg/m2 | 24.59 (3.84) | 23.91 (4.49) | 24.23 (4.16)
Neo-adjuvant chemotherapy [Count of Participants; unit: Participants] — Received neo-adjuvant chemotherapy before surgery
  Participants | 5 | 9 | 14

OUTCOME MEASURES:

1. Primary Outcome: Seroma Formation
Description: Every day for 7 days post operative period, fluid from drains was recorded (ml) daily. After discharge during follow up period, seroma formation was observed if seroma was observed, aspiration was performed and recorded.
Time Frame: Every day for 7 days post operative period and after discharge 7, 15, 21, 42, 63, 84 days during follow up period.
Population: Analysis population is patients whom randomized were performed operation as randomized and have data during follow up period.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Flap Fixation | Non Flap Fixation
Number analyzed (Participants) | 34 | 34
ml
  post operative day 0 | 54.27 (27.47) | 59.56 (49.78)
  post operative day 1 | 102.21 (40.02) | 117.94 (43.14)
  post operative day 2 | 85.00 (40.82) | 94.24 (39.06)
  post operative day 3 | 63.38 (26.90) | 82.50 (45.75)
  post operative day 4 | 53.68 (24.81) | 60.29 (29.64)
  post operative day 5 | 45.59 (23.05) | 55.00 (28.37)
  post operative day 6 | 30.59 (18.37) | 42.06 (23.36)
  post operative day 7 | 15.44 (14.27) | 26.18 (21.61)
  Follow up 7 days | 40.00 (18.26) | 86.19 (56.88)
  Follow up 15 days | 20.00 (0.00) | 72.50 (55.00)
  Follow up 21 days | 0.00 (0.00) | 72.50 (55.00)
  Follow up 42 days | 0.00 (0.00) | 86.25 (31.98)
  Follow up 63 days | 0.00 (0.00) | 30.00 (0.00)
  Follow up 84 days | 0.00 (0.00) | 0.00 (0.00)
Statistical Analysis 1: Comparison: Flap Fixation vs Non Flap Fixation; Test type: Superiority; p < 0.005, t-test, 2 sided

2. Secondary Outcome: Complication After Surgery 1. Wound Infection 2. Joint Stiffness 3. Visit Before the Appointment Date
Description: 1. wound infection; any clinical signs and symptoms of wound infection, redness , swelling, wound dehiscence, of Fever > 38 C.
  2. Joint stiffness; limitation of range of movement of Shoulder same side of mastectomy.
  3. Visit before the appointment date; any visit relevant surgical conditions before appointment.
Time Frame: Data were assessed 7 days after operation, after discharge 7 days, 15 days, 21 days, 42 days, 63 days, 84 days. Data from any time point were combined by counted and sum number of specific outcome of interest.
Measure: Count of Participants; unit: Participants
Arm/Group | Flap Fixation | Non Flap Fixation
Number analyzed (Participants) | 34 | 34
Participants
  wound infection | 0 | 2
  joint stiffness | 3 | 2
  visit before follow up date | 0 | 6
Statistical Analysis 1: Comparison: Flap Fixation vs Non Flap Fixation; Test type: Superiority; p < 0.05, Fisher Exact

ADVERSE EVENTS:
Time Frame: 3 months after operation
Description: wound infection, joint stiffness, visit before appointment
Arm/Group | Flap Fixation (n=34) | Non Flap Fixation (n=34)
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 3/34 | 10/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flap Fixation (n=34) (N=34) | Non Flap Fixation (n=34) (N=34)
Wound infection (Infections and infestations) | 0 (0) | 2 (2) — surgical wound infection, joint stiffness
Joint stiffness (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) — Limitation of movement of should joint
visit before appointment (Injury, poisoning and procedural complications) | 0 (0) | 6 (6) — any visit before appointment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-10): https://cdn.clinicaltrials.gov/large-docs/96/NCT06243796/Prot_SAP_000.pdf